CLINICAL TRIAL: NCT05959174
Title: Development of Algorithm for 3d Printed Michigan Appliances in Patients With Temporomandibular Disorders
Brief Title: Evaluation of 3D Michigan Appliance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofacial surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Myofacial Pain Syndromes
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3d printed appliance (Active Comparator)
  Interventions: Device: 3D printed mitchigen appliance
- side chair appliance (Active Comparator)
  Interventions: Device: side chair appliance

INTERVENTIONS:
Device: 3D printed mitchigen appliance — the process of appliance construction done by intra-oral scanning of the arch and 3d printing
  Arms: 3d printed appliance
Device: side chair appliance — the impresion will be taken to make a cast to reconstruct the appliance
  Arms: side chair appliance

SUMMARY:
* 20 patients will be divided into 2 groups
* Group 1 : in which conventional appliance will be constructed after alginate impression
* Group 2 : in which 3d printed appliance will be constructed after intra-oral scanning

ELIGIBILITY:
Inclusion Criteria:

* Patient with bruxism
* Trigger points
* Medically stable

Exclusion Criteria:

* • absence of other TMJ problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | Change from immediate postoperative to 6 months
  pain assessment by visual analog scale (0-10) as 0 means no pain and 10 means severe pain immediately postoperative and 6 months later

CONTACTS AND LOCATIONS:
Locations (1):
- Shaimaa Refahee, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided